CLINICAL TRIAL: NCT03527797
Title: Diaphragm-protective Mechanical Ventilation in Critically Ill Patients: A Randomized Controlled Pilot Study
Brief Title: Diaphragm Protective Ventilation in the Intensive Care Unit
Acronym: DiaPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof.dr. L.M.A. Heunks, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL62486.029.17
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Critical Illness; Muscle Weakness; Muscle Damage; Respiration, Artificial; Respiratory, Diaphragm
Keywords: Critical illness associated diaphragm weakness; Mechanical ventilation; Critical illness; Respiratory muscle dysfunction
MeSH Terms: conditions — Critical Illness; Muscle Weakness; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care
- Intervention (Experimental): Titration of support level
  Interventions: Other: Titration of support level

INTERVENTIONS:
Other: Titration of support level — Increasing support in case diaphragm activity is too high. Decreasing support in case diaphragm activity is too low.
  Arms: Intervention

SUMMARY:
Due to an accident, pneumonia or surgery, patients can have severe shortness of breath or lung damage to such an extent that it compromises vital functions. At such times, mechanical ventilation can be lifesaving. The ventilator temporarily takes over the function of the respiratory muscles to ensure adequate uptake of oxygen and removal of carbon dioxide. Mechanical ventilation can usually be stopped quickly after the initial disease has been treated. Unfortunately, in up to 25-40% of ventilated patients it takes several days to weeks before mechanical ventilation can be discontinued, even after treatment of the initial disease. This phenomenon is termed weaning failure. Weakness of the respiratory muscles, such as the diaphragm, is one of the leading causes of weaning failure.

Like other skeletal muscles, the diaphragm can become weakened if it is used too little. This happens often during mechanical ventilation because of excessive assistance provided by the ventilator or use of sedative medication. Excessive activity of the diaphragm can also lead to damage and weakness, just like in other muscles that have to perform excessive amounts for a prolonged period of time. Additionally, excessive work by the diaphragm might have a direct damaging effect on the lungs, which leads to a vicious cycle. As such, it is very important to find a balance between resting the diaphragm (which may lead to weakness) and placing excessive work on the diaphragm (which can damage the diaphragm and possibly the lungs).

In this study, the investigators want to test whether insufficient activity and excessive activity of the diaphragm during mechanical ventilation can be prevented or reduced. The investigators plan to measure the diaphragm activity in 40 participants on mechanical ventilation. Participants will be randomly assigned to the intervention group or the control group. In the intervention group, ventilator support levels will be adjusted according to the observed diaphragm activity, in an attempt to ensure adequate diaphragm activity. The control group receives usual care. The hypothesis is that adjusting the level of support provided by the ventilator is a feasible method to improve the time that the diaphragm operates within acceptable levels of activity over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Receives partially supported mechanical ventilation
* Estimated duration of mechanical ventilation after inclusion of at least 24 hours, as estimated by the attending physician

Exclusion Criteria:

* Known neuromuscular disease
* Contra-indications for nasogastric intubation (upper airway surgery, bleeding disorders)
* Expected difficulties in obtaining reliable pressure measurements, such as known airleak into pleural space or diaphragmatic herniation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Adequate diaphragm loading | 24 hours
  Percentage of time that the diaphragm operates within physiological levels of activity (Transdiaphragmatic pressure per breath between 3-12 cmH2O).

SECONDARY OUTCOMES:
Pressure-time product of diaphragm activity | 24 hours
  Average pressure-time product of the diaphragm calculated as the time-integral of transdiaphragmatic pressure, reported and compared between intervention and control
Work of breathing | 24 hours
  Average work per breath and work per minute, calculated as the volume-pressure integral of esophageal pressure, reported and compared between intervention and control
Markers for lung-protective ventilation | 24 hours
  Average transpulmonary pressure, tidal volumes, plateau airway pressures, markers for systemic inflammation and mechanical power reported and compared between intervention and control
Patient ventilator interaction | 24 hours
  Average percentage of asynchrony events, calculated as number of asynchronies / total breathing cycles * 100%, reported and compared between intervention and control

CONTACTS AND LOCATIONS:
Overall Officials: Leo M Heunks, MD, PhD, Principal Investigator — Professor of Experimental Intensive Care; Angélique Spoelstra - de Man, MD, PhD, Study Chair — Intensivist
Locations (1):
- VU University medical center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided